CLINICAL TRIAL: NCT01069575
Title: Phase I Study of Cancer Vaccine Therapy Using Epitope Peptide Restricted to HLA-A*24 (URLC10,CDCA1,KIF20A) in Patients With Non-small Cell Lung Cancer Refractory to Standard Therapy
Brief Title: Safety Study of Peptide Cancer Vaccine To Treat HLA-A*24-positive Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shiga University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Principal Investigator, Yataro Daigo, Professor, Director of Cancer Center, Shiga University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUMS-21-72; UMIN000003189 (Other: UMIN)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: URLC10; CDCA1; KIF20A; lung cancer; vaccine; HLA-A*2402
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — NUF2 protein, human; LY6K protein, human; KIF20A protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- URLC10-CDCA1-KIF20A 1mg (Experimental): Patients will be vaccinated once a week for four weeks of a treatment cycle. On each vaccination day, the HLA-A*2402-restricted URLC10 peptide (1mg), CDCA1 peptide (1mg) and KIF20A peptide(1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection.
  Interventions: Biological: HLA-A*2402restricted URLC10, CDCA1, and KIF20A peptides
- URLC10-CDCA1-KIF20A 2mg (Experimental): Patients will be vaccinated once a week for four weeks of a treatment cycle. On each vaccination day, the HLA-A*2402-restricted URLC10 peptide (2mg), CDCA1 peptide (2mg) and KIF20A peptide(2mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection.
  Interventions: Biological: HLA-A*2402restricted URLC10, CDCA1, and KIF20A peptides
- URLC10-CDCA1-KIF20A 3mg (Experimental): Patients will be vaccinated once a week for four weeks of a treatment cycle. On each vaccination day, the HLA-A*2402-restricted URLC10 peptide (3mg), CDCA1 peptide (3mg) and KIF20A peptide(3mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection.
  Interventions: Biological: HLA-A*2402restricted URLC10, CDCA1, and KIF20A peptides

INTERVENTIONS:
Biological: HLA-A*2402restricted URLC10, CDCA1, and KIF20A peptides — Escalating doses of every peptide will be administered by subcutaneous injection on days 1, 8, 15 and 22 of each treatment cycle. Planned doses of peptides are 1.0mg, 2.0mg and 3.0mg.
  Other Names: URLC10, CDCA1, and KIF20A

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, immune response and clinical efficacies of HLA-A*2402 restricted epitope peptides URLC10, CDCA1, and KIF20A emulsified with Montanide ISA 51 for advanced non-small cell lung cancers.

DETAILED DESCRIPTION:
The investigators previously identified three novel HLA-A*2402-restricted epitope peptides, which were derived from three cancer-testis antigens, URLC10, CDCA1, and KIF20A, as targets for cancer vaccination against lung cancer. In this phase I trial, the investigators examine using a combination of these three peptides the safety, immunogenicity, and antitumor effect of vaccine treatment for HLA-A*2402-positive advanced non-small cell lung cancer patients who failed to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. NSCLC that can not undergo curative surgery and treatment, and is refractory to standard chemotherapy and radiotherapy
2. ECOG performance status 0-2
3. Age between 20 to 85
4. Clinical efficacy can be evaluated by some methods
5. No prior chemotherapy, radiation therapy, hyperthermia or immunotherapy within 4 weeks
6. Life expectancy > 3 months
7. Laboratory values as follows 1500/mm3 < WBC < 15000/mm3 Platelet count > 75000/mm3 Asparate transaminase < 3 X cutoff value Alanine transaminase < 3 X cutoff value Total bilirubin < 3 X cutoff value Serum creatinine < 2X cutoff value
8. HLA-A*2402
9. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Active and uncontrolled cardiac disease (i.e. coronary syndromes, arrhythmia)
2. Myocardial infarction within six months before entry
3. Breastfeeding and Pregnancy (woman of child bearing potential)
4. Active and uncontrolled infectious disease
5. Concurrent treatment with steroids or immunosuppressing agent
6. Other malignancy requiring treatment
7. Non-cured traumatic wound
8. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-02; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety (NCI CTCAE version3): the number of adverse events of vaccination therapy. | 2 months
Evaluation of tolerability (maximum tolerated dose, MTD and dose limiting toxicity, DLT) for the determination of the recommended dose for next phase trial. | 2 months

SECONDARY OUTCOMES:
Immunological responses including peptides specific CTL, antigen cascade, regulatory T cells, cancer antigens and HLA levels | 2 months (every time point(s) at which each course is completed)
Evaluation of clinical efficacy: Objective response rate (RECIST1.1), Tumor markers, Overall survival, Progression free survival. | 2 months (every time point(s) at which each course is completed)

CONTACTS AND LOCATIONS:
Overall Officials: Yataro Daigo, MD, PhD, Principal Investigator — Department of Medical Oncology, Shiga University of Medical Science
Locations (1):
- Shiga University of Medical Science Hospital, Ōtsu, Shiga, Japan

REFERENCES:
- [Background] Kono K, Mizukami Y, Daigo Y, Takano A, Masuda K, Yoshida K, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Vaccination with multiple peptides derived from novel cancer-testis antigens can induce specific T-cell responses and clinical responses in advanced esophageal cancer. Cancer Sci. 2009 Aug;100(8):1502-9. doi: 10.1111/j.1349-7006.2009.01200.x. Epub 2009 May 14. PMID 19459850
- [Background] Harao M, Hirata S, Irie A, Senju S, Nakatsura T, Komori H, Ikuta Y, Yokomine K, Imai K, Inoue M, Harada K, Mori T, Tsunoda T, Nakatsuru S, Daigo Y, Nomori H, Nakamura Y, Baba H, Nishimura Y. HLA-A2-restricted CTL epitopes of a novel lung cancer-associated cancer testis antigen, cell division cycle associated 1, can induce tumor-reactive CTL. Int J Cancer. 2008 Dec 1;123(11):2616-25. doi: 10.1002/ijc.23823. PMID 18770861
- [Background] Mizukami Y, Kono K, Daigo Y, Takano A, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Detection of novel cancer-testis antigen-specific T-cell responses in TIL, regional lymph nodes, and PBL in patients with esophageal squamous cell carcinoma. Cancer Sci. 2008 Jul;99(7):1448-54. doi: 10.1111/j.1349-7006.2008.00844.x. Epub 2008 Apr 30. PMID 18452554
- [Background] Daigo Y, Nakamura Y. From cancer genomics to thoracic oncology: discovery of new biomarkers and therapeutic targets for lung and esophageal carcinoma. Gen Thorac Cardiovasc Surg. 2008 Feb;56(2):43-53. doi: 10.1007/s11748-007-0211-x. Epub 2008 Feb 24. PMID 18297458
- [Background] Ishikawa N, Takano A, Yasui W, Inai K, Nishimura H, Ito H, Miyagi Y, Nakayama H, Fujita M, Hosokawa M, Tsuchiya E, Kohno N, Nakamura Y, Daigo Y. Cancer-testis antigen lymphocyte antigen 6 complex locus K is a serologic biomarker and a therapeutic target for lung and esophageal carcinomas. Cancer Res. 2007 Dec 15;67(24):11601-11. doi: 10.1158/0008-5472.CAN-07-3243. PMID 18089789
- [Background] Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci. 2007 Nov;98(11):1803-8. doi: 10.1111/j.1349-7006.2007.00603.x. PMID 17784873
- [Background] Hayama S, Daigo Y, Kato T, Ishikawa N, Yamabuki T, Miyamoto M, Ito T, Tsuchiya E, Kondo S, Nakamura Y. Activation of CDCA1-KNTC2, members of centromere protein complex, involved in pulmonary carcinogenesis. Cancer Res. 2006 Nov 1;66(21):10339-48. doi: 10.1158/0008-5472.CAN-06-2137. PMID 17079454